CLINICAL TRIAL: NCT04598672
Title: Cognitive Behavioral Therapy for Insomnia (CBTi) in Patients With Somatic Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Responsible Party: Principal Investigator, Kåre Osnes, Principal investigator, Diakonhjemmet Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017/516 (PVO OUS)
Record Dates: First submitted 2020-07-06; First posted 2020-10-22 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Insomnia; Insomnia Chronic; Sleep Initiation and Maintenance Disorders; Sleep Disorder; Sleep Disturbance; Chronic Disease; Insomnia Due to Medical Condition; Insomnia, Psychophysiological
Keywords: Insomnia; Insomnia and co-morbid somatic disease; Cognitive behavioral therapy for insomnia; CBTi
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders; Parasomnias; Chronic Disease | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive behavioral therapy for insomnia (CBTi) (Experimental)
  Interventions: Behavioral: Cognitive behavioral therapy for insomnia (CBTi)

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy for insomnia (CBTi) — Patients will undergo a 7 sessions course in cognitive behavioral therapy for insomnia.

SUMMARY:
Insomnia is common with co-morbid somatic disease, e.g. rheumatic disease, cancer, heart and lung disease or gastrointestinal disorders. Pain, breathing difficulties and other symptoms of disease can worsen sleep problems and cause insomnia. In turn, insomnia may aggravate pain, fatigue and reduce quality of life in patients with somatic disorders. This project aims to evaluate a course offered to patients with insomnia and somatic disease at Diakonhjemmet Hospital. The course is based on cognitive behavioral therapy, a documented treatment for insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years with insomnia and co-morbid somatic disease.

Exclusion Criteria:

* Unable to provide informed consent
* Unable to read and/or understand Norwegian
* Unable to complete a survey
* Severe mental disorder, e.g. schizophrenia and bipolar disorder
* Mental retardation or dementia
* Known substance abuse
* Sleep disorders, e.g. narcolepsy or hypersomnia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in severity of insomnia | At baseline (before first session), at session 6 (last ordinary session, 5-7 weeks after baseline), at session 7 (2 months after last ordinary session) and 6 months after completing the course.
  All patients included in the study will be asked to complete the Insomnia Severity Index (ISI; Minimum value = 0; Maximum value = 4. Higher scores mean worse outcome) to assess for any changes in symptoms of insomnia.
Change in symptoms of insomnia | At baseline (before first session), at session 6 (last ordinary session, 5-7 weeks after baseline), at session 7 (2 months after last ordinary session) and 6 months after completing the course.
  All patients included in the study will be asked to complete the Bergen Insomnia Scale ( Minimum value = 0; Maximum value = 7. Higher scores mean worse outcome) to assess for any changes in symptoms of insomnia

SECONDARY OUTCOMES:
Change in sleep efficiency | Calculations of sleep efficiency at baseline (before first session), at session 6 (last ordinary session, 5-7 weeks after baseline), at session 7 (2 months after last ordinary session) and 6 months after completing the course, will be compared.
  All patients included in the study will be asked to keep at sleep diary for the whole duration of the course. Sleep efficiency will be calculated based on the sleep diary.
Change in dysfunctional beliefs and attitudes about sleep | At baseline (before first session), at session 6 (last ordinary session, 5-7 weeks after baseline), at session 7 (2 months after last ordinary session) and 6 months after completing the course.
  All patients included in the study will be asked to complete the Dysfunctional Beliefs and Attitudes about Sleep scale (DBAS-16; Minimum = 0; Maximum = 10. Higher values mean worse outcome) to assess for any changes in dysfunctional beliefs and attitudes about sleep.
Change in daytime rumination about tiredness and negative consequences of lack of sleep | At baseline (before first session), at session 6 (last ordinary session, 5-7 weeks after baseline), at session 7 (2 months after last ordinary session) and 6 months after completing the course.
  All patients included in the study will be asked to complete the Daytime Insomnia Symptom Response Scale (DISRS; Minimum = 1; Maximum = 4. Higher values mean worse outcome) to assess for any changes in rumination about insomnia symptoms.
Change in compliance with sleep hygiene measures | At baseline (before first session), at session 6 (last ordinary session, 5-7 weeks after baseline), at session 7 (2 months after last ordinary session) and 6 months after completing the course.
  All patients included in the study will be asked to complete the Sleep Hygiene Index (SHI-13; Minimum value = 1; Maximum value = 5. Higher values mean worse outcome) to assess for any changes in compliance with sleep hygiene measures.
Change in symptoms of depression | At baseline (before first session), at session 6 (last ordinary session, 5-7 weeks after baseline), at session 7 (2 months after last ordinary session) and 6 months after completing the course.]
  All patients included in the study will be asked to complete the Patient Health Questionnaire-9 (PHQ-9; Minimum value = 0; Maximum value = 3. Higher values mean worse outcome) to assess for any changes in symptoms of depression.
Change in symptoms of anxiety | At baseline (before first session), at session 6 (last ordinary session, 5-7 weeks after baseline), at session 7 (2 months after last ordinary session) and 6 months after completing the course
  All patients included in the study will be asked to complete the Generalized Anxiety Disorder Scale-7 (GAD-7; Minimum value = 0; Maximum value = 3. Higher values mean worse outcome) to assess for any changes in symptoms of anxiety.
Change in somatic symptoms | At baseline (before first session), at session 6 (last ordinary session, 5-7 weeks after baseline), at session 7 (2 months after last ordinary session) and 6 months after completing the course
  All patients included in the study will be asked to complete the Somatic Symptom Scale-9 (SSS-8; Minimum value = 0; Maximum value = 4. Higher value mean worse outcome) to assess for any changes in somatic symptom burden

CONTACTS AND LOCATIONS:
Overall Officials: Kåre Osnes, M.D., Ph.D., Principal Investigator — Department of Psychiatry, Diakonhjemmet Hospital, Oslo, Norway
Locations (1):
- Department of Psychiatry, Diakonhjemmet Hospital, Oslo, Norway, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No